CLINICAL TRIAL: NCT06837662
Title: Designing Intensive Primary Care Interventions to Improve Addiction Treatment for Medically and Socially Complex Patients: The "MOUD PLUS (MOUD+)" Study
Brief Title: The MOUD Plus Pilot: Counseling and Peer Support to Support Retention for Medically Complex Patients With Opioid Use Disorder Seen In Primary Care
Acronym: MOUD+
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Central City Concern (Unknown)
Responsible Party: Principal Investigator, Brian L Chan, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STUDY00024006; 5K23DA053390 (NIH)
Record Dates: First submitted 2025-02-14; First posted 2025-02-20 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Opioid Dependence; Substance Abuse Disorders; Complex Medical Patients; Primary Care Patients With Chronic Conditions
Keywords: opioid use disorder; medications for opioid use disorder; recovery capital; collaborative care model; addiction treatment
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Therapeutics; Primary Health Care

STUDY DESIGN:
Intervention Model Description: "MOUD Plus": New Components to support OUD and medical complexity
  1. Engagement with an Integrated Substance Use Disorders (SUDS) Counselor for medical complexity to aid in rapport building, brief counseling interventions (e.g., motivational interviewing, harm reduction counseling), and care coordination.
  2. Referral and coordination with outside peer organizations that work with the program to assist medically complex clients to support self-efficacy and treatment goals.
  3. Enhanced care coordination and panel management to address continuity of care and medication management for those enrolled.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Care providers may be masked to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MOUD Plus Arm (treatment as usual + integrated counseling and peer referral) (Experimental): Treatment as usual (prescriber trained in low threshold MOUD prescribing practices) plus coordinated warm-handoffs with integrated counseling services and coordinated referral to community based peer services
  Interventions: Behavioral: MOUD "Plus" Intervention (treatment as usual + coordinated counseling and referral to community based peer)
- Treatment as usual Arm (low threshold MOUD prescribing in primary care) (Active Comparator): Current treatment as usual consists of scheduled appointments with prescribers who are trained in low-threshold MOUD prescribing practices and who are part of a patient centered medical home model of care
  Interventions: Behavioral: Treatment As Usual (primary care with low threshold MOUD prescribing)

INTERVENTIONS:
Behavioral: MOUD "Plus" Intervention (treatment as usual + coordinated counseling and referral to community based peer) — In addition to treatment as usual (clinic visits for primary care and MOUD), patients will meet with clinic based addictions counselor who provides 1) rapport building ; 2) brief counseling interventions (e.g. motivational interviewing, change talk/solutions based therapy, harm reduction counseling); 3) referral to community resources. Patients will also be referred to community based peer recovery services who are credentialed and trained to "meet the person where they are" in the community and provide advocacy and support for client directed goals.
  Other Names: collaborative care; integrated behavioral health; MOUD Plus
  Arms: MOUD Plus Arm (treatment as usual + integrated counseling and peer referral)
Behavioral: Treatment As Usual (primary care with low threshold MOUD prescribing) — Treatment as usual arm consists of primary care clinical appointments with prescribers who treat medical issues and are trained to diagnosis and treat OUD using low threshold prescribing approaches.
  Other Names: usual care; treatment as usual; low-threshold MOUD prescribing
  Arms: Treatment as usual Arm (low threshold MOUD prescribing in primary care)

SUMMARY:
The goal of this pilot clinical trial is to learn if a community informed designed program of addiction counseling with coordinated community peer navigator for people with Opioid Use Disorder (OUD) and other medical conditions can improve engagement in primary care and retention on buprenorphine.

The main questions it aims to answer are:

* Does the addition of a counseling and peer referral interventions in addition to usual primary care with low-threshold buprenorphine increase retention on medications for opioid use disorder?
* Does the addition of counseling and peer referral intervention in addition to usual primary care with low-threshold buprenorphine increase engagement in primary care?

Researchers will compare the MOUD "Plus" intervention compared to primary care treatment as usual low-threshold buprenorphine prescribing practice to see if MOUD "Plus" improves retention and engagement.

Participants will upon screening and enrollment:

* Meet with prescribers who will determine dose of buprenorphine and assess other medical issues as per treatment as usual with visits every 2-4 weeks
* Meet with the integrated addictions counselor to develop rapport and support around clinic engagement, brief counseling intervention, and coordination of care in support of their MOUD
* Be referred to a community based peer who meets with participants outside the clinic for support and advocacy for patient directed recovery goals
* Meet with the research coordinator at 2, 3, and 6 months to complete follow-up surveys about their care and experiences

DETAILED DESCRIPTION:
This is a pilot randomized controlled trial (N=70) comparing the refined team-based collaborative care model ("MOUD Plus") to treatment as usual.

The hypothesis is that this team-based intervention, called "MOUD-Plus", consisting of prescribers along with integrated substance use counselor, and referral to community based peer recovery support, can improve care engagement and retention on MOUD by increasing engagement, building trust, and offering patient directed therapeutic and peer-enhanced support for their treatment on MOUD.

Main existing components of MOUD: ("Treatment as Usual")

1. Scheduled or Walk in clinic M-F 8-5 pm
2. Visits with buprenorphine waivered prescriber
3. Prescribers are trained to initiate and continue treatment same day ("low threshold" prescribing)
4. Connection to usual primary care services
5. On-site lab, pharmacy, and screening for HIV, hep C with referral to treatment

"MOUD Plus": New Components to support OUD and medical complexity

1. Engagement with an Integrated Substance Use Disorders (SUDS) Counselor for medical complexity to aid in rapport building, brief counseling interventions (e.g., motivational interviewing, harm reduction counseling), and care coordination.
2. Referral and coordination with outside peer organizations that work with the program to assist medically complex clients to support self-efficacy and treatment goals.
3. Enhanced care coordination and panel management to address continuity of care and medication management for those enrolled.

Outcomes:

1. Retention on medication for opioid use disorder (MOUD) at 2, 3-months (primary), and 6-months
2. Engagement with care teams at 2, 3, and 6-months (secondary, mechanism of action)
3. Change in trust in care team, and recovery capital at 2 months, 3, and 6-months (secondary outcomes)
4. Assess feasibility, acceptability, and potential scalability of the program using the RE-AIM-QuEST framework

ELIGIBILITY:
Inclusion Criteria:

* Eligibility/Inclusion Criteria. For Aim 3, criteria we seek to recruit include:
* Patient participants 18 years and older
* Have an OUD-related diagnosis (e.g. Opioid Use Disorder in remission, Opioid Dependence, Opioid Abuse, Substance Use Disorder - opioids, etc.), or have used fentanyl or heroin over the past 30 days
* Who meet at least one of the following criteria:

  * Present to primary care at Central City Concern (CCC) within 8 weeks of starting or re-starting a treatment episode (defined as starting MOUD after not having received prescribed MOUD in an outpatient setting for OUD in the prior 30 days).
  * Who present to primary care at CCC and are not seeking treatment with MOUD and have not engaged in counseling services (e.g. harm reduction counseling) in the prior 30 days
  * Have been receiving MOUD in prior 30 days but had a return to use (used fentanyl or heroin) within the past 30 days
* Medical complexity (e.g. self-reported or verified in patient's electronic health record)
* Have access to phone and/or computer for follow-up activities
* Desire to engage in counseling and/or peer services

Exclusion Criteria:

* Patient participants who present for addiction treatment but are ineligible to receive on-going services at Central City (i.e. they have existing primary care at another location, or are currently receiving opioid use disorder treatment at another clinic, such as methadone clinic) may not participate in the study.
* Patient participants who are not able to verbally consent may not participate in the study.
* Patients who do not have addiction to opioids may not participate in the study.
* Patients who participated in Aim 2 would not be eligible for Aim 3
* Patients who lack stable phone access may not participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2026-03-21 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Retention on MOUD | assessed at 2 month, 3 months, and 6 month post enrollment
  Retention is defined as a composite measure assessed at follow-up on whether they report being prescribed and taking MOUD, and how days since the last follow-up they have been on MOUD, confirmed by chart review.

SECONDARY OUTCOMES:
Engagement with care team | Assessed at 3-month follow-up post enrollment
  Engagement with care team is defined by number of unique contacts (in person visits, telephone visits, telephone outreach, peer engagements) the participant has with each arm during the course of the study
Change in recovery capital instrument (BARC-10) | Change between baseline and assessed at 2-month, 3-month, and 6-month follow up
  We assess recovery capital using the brief assessment of recovery capital (BARC-10) which ranges from minimum of 10 to maximum of 60.
Change in patient reported trust in care team | Change between baseline and assessed at 2-month, 3-month, and 6-month follow up
  We assess trust in care team using a modified version Wake Forest Physician Trust scale which ranges from minimum of 10 to maximum of 50.

OTHER OUTCOMES:
Change in opioid use based on self-report | Baseline, 2, 3, and 6 months
  Modified Timeline Followback survey questions assess use of opioids since last time period
Change in other drug use (alcohol, methamphetamine) based on self-report | Baseline, 2, 3, and 6 months
  Modified Timeline Followback survey questions assess use of other drug use since last time period
Hospitalization and ED visits for substance use related problem | Baseline, 2, 3, and 6 months
  Patient reported survey question confirmed with medical chart review of number of hospitalizations, ED visits, or withdrawal management visits during follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Chan, MD MPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- Central City Concern, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
After completion of the study, analysis, and publication, a de-identified IPD that underlie results in a publication will be made available upon reasonable request.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Starting after publication of the main results, and for 5 years after.
Access Criteria: Anyone who makes a reasonable request to the primary investigator via email with rationale and data analysis plan/question